CLINICAL TRIAL: NCT03548415
Title: A Double-Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability, and Efficacy of ISIS 766720 (IONIS-GHR-LRx, an Antisense Inhibitor of the Growth Hormone Receptor) Administered Once Every 28 Days for 16 Weeks in Patients With Acromegaly Being Treated With Long-acting Somatostatin Receptor Ligands (SRL)
Brief Title: Safety, Tolerability, and Efficacy of IONIS-GHR-LRx in Participants With Acromegaly Being Treated With Long-acting Somatostatin Receptor Ligands
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 766720-CS2; 2017-004259-22 (EudraCT Number)
Record Dates: First submitted 2018-05-22; First posted 2018-06-07 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Acromegaly
Keywords: Acromegaly, IONIS-GHR-LRx
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received placebo by subcutaneous injection (SC) once every 4 weeks for 16 weeks.
  Interventions: Drug: Placebo
- Cohort A: IONIS GHR-LRx, 60 mg (Experimental): Participants received IONIS GHR-LRx, 60 milligrams (mg), SC, once every 4 weeks for 16 weeks.
  Interventions: Drug: IONIS-GHR-LRx
- Cohort B: IONIS GHR-LRx, 80 mg (Experimental): Participants received IONIS GHR-LRx, 80 mg, SC, once every 4 weeks for 16 weeks.
  Interventions: Drug: IONIS-GHR-LRx
- Cohort C: IONIS GHR-LRx, 120 mg (Experimental): Participants received IONIS GHR-LRx, 120 mg, SC, once every 4 weeks for 16 weeks.
  Interventions: Drug: IONIS-GHR-LRx
- Cohort D: IONIS GHR-LRx, 160 mg (Experimental): Participants received IONIS GHR-LRx, 160 mg, SC, once every 4 weeks for 16 weeks.
  Interventions: Drug: IONIS-GHR-LRx

INTERVENTIONS:
Drug: IONIS-GHR-LRx — IONIS GHR-LRx administered subcutaneously.
  Arms: Cohort A: IONIS GHR-LRx, 60 mg; Cohort B: IONIS GHR-LRx, 80 mg; Cohort C: IONIS GHR-LRx, 120 mg; Cohort D: IONIS GHR-LRx, 160 mg
Drug: Placebo — Placebo administered subcutaneously.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and efficacy of IONIS-GHR-LRx in up to 60 participants with acromegaly.

DETAILED DESCRIPTION:
This short-term study assessed changes in serum insulin-like growth factor 1 (IGF-1) over a 16-week treatment period in a participant population diagnosed with acromegaly being treated with long-acting somatostatin receptor ligands (SRL).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with documented diagnosis of acromegaly, aged 18-75 years old (inclusive) at the time of informed consent
2. Participants must be on stable maximum or maximally tolerated dose of SRL (Lanreotide Autogel or Octreotide LAR, per treating physician judgment) every 28 days for a minimum of 3 months prior to screening and will be required to continue their stable dose of SRL throughout the study. Prior use of other medications for treating acromegaly is allowed but not within 6 weeks of screening.
3. At Screening, serum insulin-like growth factor 1 (IGF-1) (performed at central lab) between 1.3 to 5 x upper limit of normal (ULN), inclusive, adjusted for age and sex
4. Females must be non-pregnant and non-lactating, and either surgically sterile, post-menopausal, abstinent, or using 1 highly effective method of birth control

Exclusion Criteria:

1. Participants who received surgery for pituitary adenoma within the last 6 months before the trial, or planning to receive surgery during the trial
2. Participants who received radiotherapy for pituitary adenoma within the last 3 years before the trial, and/or planning to receive radiotherapy during the trial
3. Participants with pituitary tumor that, per Investigator judgement, is worsening as assessed by pituitary/sellar magnetic resonance imaging (MRI) protocol at Screen or within 6 months of screening
4. Evidence of decompensated cardiac function per medical judgement and/or New York Heart Association (NYHA) class 3 or 4
5. Clinical evidence of symptomatic hyperprolactinemia that would necessitate treatment
6. Participants may not have chronic systemic use of glucocorticoids, weight loss medications or participate in weight loss programs within 2 months before randomization and during study participation.
7. Participants on anti-diabetes medication or estrogen containing medications must be on a stable dose and regimen for >= 3 months prior to screening and throughout the trial
8. Participants taking glucagon-like peptide 1 (GLP-1) agonists or insulin can be allowed with prior consultation with the Sponsor Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (6):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Northwestern University, Chicago, Illinois
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University (OHSU), Portland, Oregon
- Hungary (3):
  - Magyar Honvedseg Allami Egeszsegugyi Kozpont, II. sz Belgyogyaszat Osztaly, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szeged University - Szent-Gyorgyi Albert Clinical Center - I. Belgyógyászati Klinika (Internal Medicine), Szeged
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences (LSMU) Kauno klinikos - Hospital of Oncology, Kaunas
  - Vaidoto Urbanaviciaus Individuali imone - Endokrinologijos klinika, Vilnius
- Poland (6):
  - B_Serwis Popenda Sp. J. Specjalistyczna Przychodnia Lekarsk, Chorzów
  - Uniwersyteckie Centrum Kliniczne im. Prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o. o., Krakow
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Mazowiecki Szpital Brodnowski - Zespol Oddzialow Chorob Wewnetrznych, Endokrynologii i Diabetologii, Warsaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Sp. p., Wroclaw
- Romania (4):
  - Centrul Medical Unirea - Bucuresti, Endocrinologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj - Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
- Russia (10):
  - Multi-field Medical Clinic Anturium LLC, Barnaul
  - Interregional Clinical Diagnostic Center, Kazan'
  - Kuzbass Clinical Hospital n.a. S.V. Belyaev, Kemerovo
  - Federal State Budget Institution "National Medical Research Center of Endocrinology" of the Ministry of Healthcare of the Russian Federation, Moscow
  - I.M. Sechenov Moscow First State Medical University, Moscow
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Orenburg Regional Clinical Hospital, Endocrinology Department, Orenburg
  - Rostov State Medical University, Rostov-on-Don
  - Almazov National Medical Research Centre, Saint Petersburg
  - State Budget Healthcare Institution of the Tver Region, Tver'
- Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 24 investigative sites in Lithuania, Hungary, the United States of America, Serbia, Russia, Poland, and Romania from 13 September 2018 to 02 April 2021.
Pre-assignment Details: Adult participants diagnosed with acromegaly were randomized into 4 cohorts [Cohorts A and B in 2:1 ratio; Cohorts C and D in 5:1 ratio] to receive IONIS GHR-LRx or placebo. Due to enrollment difficulties associated with (COVID-19) pandemic, treatment groups IONIS GHR-LRx, 120 mg and IONIS GHR-LRx, 160 mg did not complete enrollment resulting in cohort sizes smaller than planned.
Period: Overall Study
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg
Started | 12 | 12 | 11 | 2 | 6
Per-Protocol Set (The Per-Protocol Set included all randomized participants who received at least 5 of the 6 doses of Study Drug and had at least one post-baseline efficacy or pharmacodynamic assessment, with the first 3 doses administered on schedule, and had no significant protocol deviations that would have been expected to affect efficacy.) | 12 | 11 | 11 | 2 | 5
Completed | 12 | 11 | 11 | 2 | 5
Not Completed | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event or Serious Adverse Event | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who were randomized and received at least one dose of Study Drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg | Total
Number analyzed (Participants) | 12 | 12 | 11 | 2 | 6 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (11.7) | 48.9 (13.6) | 52.1 (14.9) | 53.5 (2.1) | 46.0 (13.3) | 48.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 0 | 4 | 27
  Male | 4 | 3 | 5 | 2 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 11 | 2 | 6 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 00 | 1 | 1
  White | 12 | 12 | 11 | 2 | 5 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum Insulin-like Growth Factor-1 (IGF-1) From Baseline to 28 Days After Last Dose
Description: IGF-1 is a hormone that manages the effects of growth hormone (GH) in the body. Percent change from Baseline in IGF-1 levels was measured at Day 141. Baseline was defined as the last non-missing value prior to the first administration of Study Drug (ISIS 766720 or placebo). A negative percent change from Baseline indicated improvement. To perform a meaningful assessment of the pharmacodynamic (PD) activity of ISIS 766720, the lower dose groups (60 mg and 80 mg) and higher dose groups (120 mg and 160 mg) were combined to achieve group size of 7 or more for PD assessments and these were designated as low-dose and high-dose groups respectively.
Time Frame: Baseline and 28 days after last dose (Day 141)
Population: The Per-protocol Set included all randomized participants who received at least one dose of Study Drug and had at least one post-baseline efficacy or pharmacodynamic assessment, received at least 5 of the 6 doses of Study Drug with the first 3 doses administered on schedule, and had no significant protocol deviations that would have been expected to affect efficacy. Low dose refers to 60 mg or 80 mg, High dose refers to 120 mg or 160 mg.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- ISIS 766720 Low Dose: Participants received IONIS GHR-LRx, 60 or 80 milligrams (mg), SC, once every 4 weeks for 16 weeks.
- ISIS 766720 High Dose: Participants received IONIS GHR-LRx, 120 or 160 mg, SC, once every 4 weeks for 16 weeks.
Arm/Group | Placebo | ISIS 766720 Low Dose | ISIS 766720 High Dose
Number analyzed (Participants) | 12 | 22 | 7
percent change | 8.9 (31.5) | -2.8 (33.1) | -7.5 (16.3)
Statistical Analysis 1: Comparison: Placebo vs ISIS 766720 Low Dose; Test type: Superiority; p = 0.306, Van Elteren test — The p-value was analyzed using the nonparametric test, Van Elteren test with IGF-1 level as stratification factor

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event that occurred after the initiation of study drug dosing and before the end of the follow-up period.
Time Frame: Up to 211 days
Population: The Safety Set included all participants who were randomized and received at least one dose of Study Drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg
Number analyzed (Participants) | 12 | 12 | 11 | 2 | 6
Participants | 8 | 11 | 7 | 2 | 5

3. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Vital Sign Findings
Description: Vitals signs included blood pressure, heart rate, respiratory rate, and temperature recorded throughout the study. Clinical significance was determined by the investigator.
Time Frame: Up to 211 days
Population: The Safety Set included all participants who were randomized and received at least one dose of Study Drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg
Number analyzed (Participants) | 12 | 12 | 11 | 2 | 6
Participants
  Hypotension | 0 | 1 | 0 | 0 | 0
  Hypertension | 0 | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Physical Examination Findings
Description: Physical examination included weight and body mass index (BMI) recorded throughout the study. Clinical significance was determined by the investigator.
Time Frame: Up to 211 days
Population: The Safety Set included all participants who were randomized and received at least one dose of Study Drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg
Number analyzed (Participants) | 12 | 12 | 11 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Laboratory Evaluation Findings
Description: Clinical laboratory assessments included clinical chemistry, hematology, and urinalysis. Clinically-significant abnormal laboratory values were reported as TEAEs if the results may, in the opinion of the Investigator, constitute or be associated with an AE.
Time Frame: Up to 211 days
Population: The Safety Set included all participants who were randomized and received at least one dose of Study Drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg
Number analyzed (Participants) | 12 | 12 | 11 | 2 | 6
Participants
  Blood urine present | 0 | 0 | 0 | 1 | 0
  Mean cell volume increased | 0 | 1 | 0 | 0 | 0
  Urine protein/creatinine ratio increased | 0 | 0 | 1 | 0 | 0
  Hyperglycaemia | 1 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG assessments included QT, QRS duration, PR interval, ventricular rate, QTcB, QTcF.
Time Frame: Up to 211 days
Population: The Safety Set included all participants who were randomized and received at least one dose of Study Drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg
Number analyzed (Participants) | 12 | 12 | 11 | 2 | 6
Participants | 2 | 2 | 1 | 1 | 0

7. Secondary Outcome: Number of Participants Achieving Normalized IGF-1 Levels to Within 1.2 Times of Gender and Age Limits at 28 Days After Last Dose
Description: Normalization of circulating IGF-1 is a validated marker for the treatment of acromegaly. IGF-1 assessments were based on a single serum sample taken in fasting conditions, prior to the study drug administration. Normal IGF-1 levels for a participant differ based on age and gender. Number of participants with a normal IGF-1 level which were 1.2 times within gender and age limits after 28 days of the last dose (Day 141) are presented. To perform a meaningful assessment of the pharmacodynamic activity of ISIS 766720, the lower dose groups (60 mg and 80 mg) and higher dose groups (120 mg and 160 mg) were combined to achieve group size of 7 or more for PD assessments and these were designated as low-dose and high-dose groups respectively.
Time Frame: Baseline to 28 days after last dose (Day 141)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ISIS 766720 Low Dose | ISIS 766720 High Dose
Number analyzed (Participants) | 12 | 22 | 7
Participants | 0 | 5 | 1

8. Secondary Outcome: Number of Participants Achieving Normalized IGF-1 Levels to Within 1.0 Times of Gender and Age Limits at 28 Days After Last Dose
Description: Normalization of circulating IGF-1 is a validated marker for the treatment of acromegaly. IGF-1 assessments were based on a single serum sample taken in fasting conditions, prior to the study drug administration. Normal IGF-1 levels for a participant differ based on age and gender. Number of participants with a normal IGF-1 level which were 1.0 times within gender and age limits after 28 days of the last dose (Day 141) are presented. To perform a meaningful assessment of the pharmacodynamic activity of ISIS 766720, the lower dose groups (60 mg and 80 mg) and higher dose groups (120 mg and 160 mg) were combined to achieve group size of 7 or more for PD assessments and these were designated as low-dose and high-dose groups respectively.
Time Frame: Baseline to 28 days after last dose (Day 141)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ISIS 766720 Low Dose | ISIS 766720 High Dose
Number analyzed (Participants) | 12 | 22 | 7
Participants | 0 | 2 | 0

9. Secondary Outcome: Change From Baseline in Serum IGF-1 Over Time
Description: IGF-1 is a hormone that manages the effects of GH in the body. Change from Baseline in IGF-1 levels was measured at multiple timepoints up to Day 211. Baseline was defined as the last non-missing value prior to the first administration of Study Drug (ISIS 766720 or placebo). A negative change from Baseline indicated improvement. To perform a meaningful assessment of the pharmacodynamic activity of ISIS 766720, the lower dose groups (60 mg and 80 mg) and higher dose groups (120 mg and 160 mg) were combined to achieve group size of 7 or more for PD assessments and these were designated as low-dose and high-dose groups respectively.
Time Frame: Baseline, Days 15, 29, 43, 57, 71, 85, 99, 112, 127, 141, 155, 183, and 211
Population: Per-protocol Set:all randomized participants who received at least one dose of Study Drug and had at least one post-baseline efficacy or PD assessment, received at least 5 of 6 doses of Study Drug with first 3 doses administered on schedule, and had no significant protocol deviations that would have been expected to affect efficacy. Number analyzed is the number of participants with data available at specific timepoints. Low dose refers to 60 mg or 80 mg,High dose refers to 120 mg or 160 mg.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Placebo | ISIS 766720 Low Dose | ISIS 766720 High Dose
Number analyzed (Participants) | 12 | 22 | 7
nanograms per milliliter
  Baseline | 386 (154) | 422 (214) | 419 (143)
  Change from Baseline at Day 15 | 33 (112) | -46 (108) | -10 (47)
  Change from Baseline at Day 29 | 23 (71) | -30 (140) | -68 (55)
  Change from Baseline at Day 43: number analyzed (Participants) | 12 | 21 | 7
  Change from Baseline at Day 43 | 17 (114) | -41 (142) | -88 (95)
  Change from Baseline at Day 57 | 52 (120) | -39 (147) | -74 (63)
  Change from Baseline at Day 71 | 9 (115) | -71 (163) | -78 (76)
  Change from Baseline at Day 85 | 9 (91) | -55 (136) | -90 (141)
  Change from Baseline at Day 99 | 13 (124) | -49 (104) | -104 (78)
  Change from Baseline at Day 112 | 31 (93) | -36 (100) | -61 (70)
  Change from Baseline at Day 127: number analyzed (Participants) | 12 | 21 | 7
  Change from Baseline at Day 127 | 19 (83) | -48 (133) | -74 (69)
  Change from Baseline at Day 141 | 20 (100) | -39 (140) | -48 (92)
  Change from Baseline at Day 155: number analyzed (Participants) | 8 | 20 | 3
  Change from Baseline at Day 155 | 1 (91) | -47 (144) | -98 (112)
  Change from Baseline at Day 183: number analyzed (Participants) | 8 | 18 | 3
  Change from Baseline at Day 183 | -13 (87) | -45 (155) | -15 (146)
  Change from Baseline at Day 211: number analyzed (Participants) | 8 | 17 | 2
  Change from Baseline at Day 211 | 13 (116) | -55 (161) | -92 (97)

10. Secondary Outcome: Percent Change From Baseline in Serum IGF-1 Over Time
Description: IGF-1 is a hormone that manages the effects of GH in the body. Percent change from Baseline in IGF-1 levels was measured at multiple timepoints up to Day 211. Baseline was defined as the last non-missing value prior to the first administration of Study Drug (ISIS 766720 or placebo). A negative percent change from Baseline indicated improvement. To perform a meaningful assessment of the pharmacodynamic activity of ISIS 766720, the lower dose groups (60 mg and 80 mg) and higher dose groups (120 mg and 160 mg) were combined to achieve group size of 7 or more for PD assessments and these were designated as low-dose and high-dose groups respectively.
Time Frame: Baseline, Days 15, 29, 43, 57, 71, 85, 99, 112, 127, 155, 183, and 211
Population: Per-protocol Set:all randomized participants who received at least one dose of Study Drug and had at least one post-baseline efficacy or PD assessment, received at least 5 of 6 doses of Study Drug with first 3 doses administered on schedule,and had no significant protocol deviations that would have been expected to affect efficacy. Number analyzed is number of participants with data available for analysis at specific timepoint.Low dose refers to 60 mg or 80 mg,High dose refers to 120mg or 160mg.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | ISIS 766720 Low Dose | ISIS 766720 High Dose
Number analyzed (Participants) | 12 | 22 | 7
percent change
  Percent Change from Baseline at Day 15 | 11.2 (31.3) | -6.0 (24.5) | -0.2 (11.9)
  Percent Change from Baseline at Day 29 | 9.3 (26.2) | -3.5 (30.0) | -14.8 (6.8)
  Percent Change from Baseline at Day 43: number analyzed (Participants) | 12 | 21 | 7
  Percent Change from Baseline at Day 43 | 9.6 (35.7) | -5.1 (28.4) | -18.3 (18.5)
  Percent Change from Baseline at Day 57 | 14.3 (34.5) | -3.4 (31.9) | -16.6 (11.6)
  Percent Change from Baseline at Day 71 | 8.8 (33.4) | -9.0 (42.0) | -16.5 (12.3)
  Percent Change from Baseline at Day 85 | 4.2 (27.2) | -5.6 (32.5) | -16.7 (19.4)
  Percent Change from Baseline at Day 99 | 6.6 (38.8) | -7.1 (30.1) | -25.1 (18.0)
  Percent Change from Baseline at Day 112 | 12.1 (29.8) | -4.0 (33.6) | -12.3 (9.3)
  Percent Change from Baseline at Day 127: number analyzed (Participants) | 12 | 21 | 7
  Percent Change from Baseline at Day 127 | 6.3 (19.6) | -4.7 (30.2) | -16.0 (9.0)
  Percent Change from Baseline at Day 141 | 8.9 (31.5) | -2.8 (33.1) | -7.5 (16.3)
  Percent Change from Baseline at Day 155: number analyzed (Participants) | 8 | 20 | 3
  Percent Change from Baseline at Day 155 | 4.1 (26.0) | -3.5 (32.0) | -18.1 (14.1)
  Percent Change from Baseline at Day 183: number analyzed (Participants) | 8 | 18 | 3
  Percent Change from Baseline at Day 183 | 0.1 (26.2) | -2.5 (38.7) | 1.6 (25.9)
  Percent Change from Baseline at Day 211: number analyzed (Participants) | 8 | 17 | 2
  Percent Change from Baseline at Day 211 | 2.2 (30.6) | -8.2 (32.7) | -15.6 (10.5)

ADVERSE EVENTS:
Time Frame: Up to 211 days
Description: The Safety Set included all participants who were randomized and received at least one dose of Study Drug.
Arm/Group | Placebo | Cohort A: IONIS GHR-LRx, 60 mg | Cohort B: IONIS GHR-LRx, 80 mg | Cohort C: IONIS GHR-LRx, 120 mg | Cohort D: IONIS GHR-LRx, 160 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/12 | 0/11 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 1/11 | 0/2 | 1/6
Other Adverse Events (participants affected / at risk) | 8/12 | 11/12 | 7/11 | 2/2 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Cohort A: IONIS GHR-LRx, 60 mg (N=12) | Cohort B: IONIS GHR-LRx, 80 mg (N=11) | Cohort C: IONIS GHR-LRx, 120 mg (N=2) | Cohort D: IONIS GHR-LRx, 160 mg (N=6)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Cohort A: IONIS GHR-LRx, 60 mg (N=12) | Cohort B: IONIS GHR-LRx, 80 mg (N=11) | Cohort C: IONIS GHR-LRx, 120 mg (N=2) | Cohort D: IONIS GHR-LRx, 160 mg (N=6)
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0
Mean cell volume increased (Investigations) | 0 | 1 | 0 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bundle branch block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Acromegaly (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
While no longer powered to assess the primary endpoint (% IGF- lowering at Day 141) in accordance with the protocol, the study did permit placebo-controlled evaluation of safety and efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03548415/Prot_SAP_000.pdf